CLINICAL TRIAL: NCT04005885
Title: A Clinical Comparison of Two Daily Disposable Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: EX-MKTG-100
Record Dates: First submitted 2019-07-01; First posted 2019-07-02 (Actual); Results first posted 2020-12-11 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Subjects and investigators will be masked to the study lenses - lenses will be overlabelled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- somofilcon A then stenfilcon A contact lens (Experimental): Participants were fitted with comfilcon A lens on a daily wear, reusable basis for 1 month, then randomized to wear somofilcon A daily disposable test lens for 1 week of daily wear and stenfilcon A daily disposable test lens for 1 week of daily wear.
  Interventions: Device: comfilcon A; Device: somofilcon A; Device: stenfilcon A
- stenfilcon A then somofilcon A contact lens (Experimental): Participants were fitted with comfilcon A lens on a daily wear, reusable basis for 1 month, then randomized to wear stenfilcon A daily disposable test lens for 1 week of daily wear and somofilcon A daily disposable test lens for 1 week of daily wear.
  Interventions: Device: comfilcon A; Device: somofilcon A; Device: stenfilcon A

INTERVENTIONS:
Device: comfilcon A — Contact Lens
  Other Names: Control Lens
Device: somofilcon A — daily disposable contact lens
  Other Names: somofilcon A daily disposable test lens; Test lens 1
Device: stenfilcon A — daily disposable contact lens
  Other Names: stenfilcon A daily disposable test lens; Test lens 2

SUMMARY:
This double-masked, randomized, bilateral, crossover, direct refit study compared the clinical performance of two daily disposable contact lenses (somofilcon A and stenfilcon A) when fitted to existing wearers of comfilcon A monthly lenses.

DETAILED DESCRIPTION:
This double-masked (subject and investigator), randomized, bilateral, crossover, direct refit study compared the clinical performance of two daily disposable test contact lenses (somofilcon A and stenfilcon A) when fitted to existing wearers of comfilcon A monthly lenses. After a month of re-useable lens wear in the comfilcon A lenses, subjects were randomized to wear each daily disposable lens type for one week.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will only be eligible for the study if:
* They are between 18 and 40 years of age (inclusive).
* They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
* They are willing and able to follow the protocol.
* They are an existing soft reusable spherical contact lens wearer in both eyes.
* They have a contact lens spherical prescription between -0.50 to -6.00D (inclusive) based on the ocular refraction.
* They have a cylindrical correction of -0.875DC or less in each eye based on the ocular refraction
* They own a wearable pair of spectacles and wear them on the day of the initial visit.
* They have distance high contrast logMAR visual acuity of 0.2 or better in each eye with their habitual spectacles.
* They agree not to participate in other clinical research for the duration of the study.

Exclusion Criteria:

* They have an ocular disorder which would normally contra-indicate contact lens wear.
* They have a systemic disorder which would normally contra-indicate contact lens wear.
* They are using any topical medication such as eye drops or ointment.
* They are aphakic.
* They have had corneal refractive surgery.
* They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
* They are pregnant or breastfeeding.
* They have any infectious disease which would, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel; or they have any immunosuppressive disease (e.g. HIV), or a history of anaphylaxis or severe allergic reaction.
* They have taken part in any other contact lens or care solution clinical trial or research, within two weeks prior to starting this study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carole Maldonado-Codina, PhD, MCOptom, FAAO, FBCLA, Principal Investigator — Eurolens Research
Locations (1):
- Eurolens Research - The University of Manchester, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects were fitted with comfilcon A for one month and then the subjects were randomized to wear two daily disposable lenses for one week.
Groups:
- Somofilcon A, Then Stenfilcon A Contact Lens: All subjects fitted with the comfilcon A lens on a daily wear, reusable basis for 1 month were randomized to wear the somofilcon A daily disposable test lens for 1 week of daily wear and stenfilcon A daily disposable test lens for 1 week of daily wear.
  comfilcon A : contact lens
  somofilcon A: daily disposable contact lens
  stenfilcon A: daily disposable contact lens
- Stenfilcon A, Then Somofilcon A Contact Lens: All subjects fitted with comfilcon A lens on a daily wear, reusable basis for 1 month were randomized to wear stenfilcon A daily disposable test lens for 1 week of daily wear and somofilcon A daily disposable test lens for 1 week of daily wear.
  comfilcon A: Contact Lens
  somofilcon A: daily disposable contact lens
  stenfilcon A: daily disposable contact lens
Period: First Intervention
Arm/Group | Somofilcon A, Then Stenfilcon A Contact Lens | Stenfilcon A, Then Somofilcon A Contact Lens
Started | 26 | 29
Completed | 25 | 28
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Second Intervention
Arm/Group | Somofilcon A, Then Stenfilcon A Contact Lens | Stenfilcon A, Then Somofilcon A Contact Lens
Started | 25 | 28
Completed | 25 | 26
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Third Intervention
Arm/Group | Somofilcon A, Then Stenfilcon A Contact Lens | Stenfilcon A, Then Somofilcon A Contact Lens
Started | 25 | 26
Completed | 25 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Subjects were randomized to wear comfilcon A lens on a daily wear, reusable basis for 1 month, then fitted and wear the somofilcon A daily disposable test lens and stenfilcon A daily disposable test lens each for 1 week of daily wear.
  comfilcon A: Contact Lens
  somofilcon A: daily disposable contact lens
  stenfilcon A: daily disposable contact lens
Arm/Group | Overall Study
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.1 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 55

OUTCOME MEASURES:

1. Primary Outcome: Subjective Scores of Comfort at Insertion After 4 Weeks of Comfilcon A Use
Description: Subjective Scores of comfort at Insertion after 4 weeks of Comfilcon A use rated on a scale 0-100 (0=causes pain, cannot be tolerated, 100=excellent, cannot be felt).
Time Frame: 4 weeks
Population: One subject discontinued after dispensing visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Comfilcon A: Participants were fitted to wear comfilcon A lens on a daily wear, reusable basis for 1 month.
  comfilcon A: Contact Lens
Arm/Group | Comfilcon A
Number analyzed (Participants) | 54
units on a scale | 89.9 (14.5)

2. Primary Outcome: Subjective Scores of Comfort on Insertion
Description: Subjective Scores of Comfort on Insertion rated on a scale 0 -100 (0=causes pain, cannot be tolerated, 100=excellent, cannot be felt).
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Somofilcon A Contact Lens: Participants were randomized to wear somofilcon A daily disposable test lens for 1 week of daily wear.
  somofilcon A: daily disposable contact lens
- Stenfilcon A Contact Lens: Participants were randomized to wear stenfilcon A daily disposable test lens for 1 week of daily wear.
  stenfilcon A: daily disposable contact lens
Arm/Group | Somofilcon A Contact Lens | Stenfilcon A Contact Lens
Number analyzed (Participants) | 51 | 52
units on a scale | 90.3 (12.6) | 90.4 (12.8)

3. Secondary Outcome: Subjective Scores on Overall Comfort After 4 Weeks of Comfilcon Use
Description: Subjective scores on overall comfort after 4 weeks of comfilcon use rated on a scale 0 -100 (0=causes pain, cannot be tolerated, 100=excellent, cannot be felt).
Time Frame: 4 weeks
Population: One Subject discontinued after dispensing visit
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Comfilcon A Contact Lens: Participants were fitted to wear comfilcon A lens on a daily wear, reusable basis for 1 month.
  comfilcon A: Contact Lens
Arm/Group | Comfilcon A Contact Lens
Number analyzed (Participants) | 54
units on a scale | 83.7 (15.5)

4. Secondary Outcome: Subjective Scores on Overall Comfort
Description: Subjective Scores on overall comfort rated on a scale 0 - 100 (0=causes pain, cannot be tolerated, 100=excellent, cannot be felt).
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A Contact Lens | Stenfilcon A Contact Lens
Number analyzed (Participants) | 51 | 52
units on a scale | 84.0 (16.8) | 85.7 (13.2)

5. Secondary Outcome: Subjective Scores on Comfort Before Removal After 4 Weeks of Comfilcon Use
Description: Subjective Scores on Comfort before removal after 4 weeks of comfilcon use rated on a scale 0-100 (0=causes pain, cannot be tolerated, 100=excellent, cannot be felt).
Time Frame: 4 weeks
Population: One Subject discontinued after dispensing visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Contact Lens
Number analyzed (Participants) | 54
units on a scale | 73.1 (20.2)

6. Secondary Outcome: Subjective Scores on Comfort Before Removal
Description: Subjective Scores on Comfort before removal rated on a scale 0-100 (0=causes pain, cannot be tolerated, 100=excellent, cannot be felt).
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A Contact Lens | Stenfilcon A Contact Lens
Number analyzed (Participants) | 51 | 52
units on a scale | 77.6 (19.0) | 79.3 (15.8)

7. Secondary Outcome: Number of Participants With Horizontal Lens Centration Grade
Description: Number of Participants with Horizontal Lens centration graded on scale of -2 to 2 ( -2= Extremely nasal, -1 slightly nasal, 0=optimum, 1=slightly temporal, 2=extremely temporal)
Time Frame: Baseline (after 5 minutes of lens dispense)
Measure: Count of Participants; unit: Participants
Arm/Group | Comfilcon A Contact Lens | Somofilcon A Contact Lens | Stenfilcon A Contact Lens
Number analyzed (Participants) | 55 | 51 | 53
Participants
  Extremely nasal | 0 | 0 | 0
  Slightly nasal | 0 | 2 | 2
  Optimum | 35 | 19 | 33
  Slightly Temporal | 20 | 30 | 18
  Extremely Temporal | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Horizontal Lens Centration Grade After 4 Weeks of Comfilcon A Wear
Description: Number of Participants with Horizontal lens centration after 4 weeks of comfilcon A wear graded on scale of -2 to 2 ( -2= Extremely nasal, -1 slightly nasal, 0=optimum, 1=slightly temporal, 2=extremely temporal)
Time Frame: 4 weeks
Population: One subject discontinued after dispensing visit
Measure: Count of Participants; unit: Participants
Arm/Group | Comfilcon A Contact Lens
Number analyzed (Participants) | 54
Participants
  Extremely nasal | 0
  Slightly nasal | 1
  Optimum | 32
  Slightly Temporal | 21
  Extremely Temporal | 0

9. Secondary Outcome: Number of Participants With Horizontal Lens Centration Grade
Description: as for outcome 7
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Contact Lens | Stenfilcon A Contact Lens
Number analyzed (Participants) | 51 | 52
Participants
  Extremely nasal | 0 | 0
  Slightly nasal | 3 | 1
  Optimum | 20 | 30
  Slightly Temporal | 28 | 21
  Extremely Temporal | 0 | 0

10. Secondary Outcome: Number of Participants With Vertical Lens Centration Grade
Description: Number of Participants with Vertical lens centration graded on a scale of -2 to 2 ( -2= Extremely inferior, -1 slightly inferior, 0=optimum, 1=slightly superior, 2=extremely superior)
Time Frame: Baseline (After 5 minutes of lens dispense)
Measure: Count of Participants; unit: Participants
Arm/Group | Comfilcon A Contact Lens | Somofilcon A Contact Lens | Stenfilcon A Contact Lens
Number analyzed (Participants) | 55 | 51 | 53
Participants
  Extremely Inferior | 0 | 0 | 0
  Slightly Inferior | 12 | 8 | 7
  Optimum | 35 | 23 | 35
  Slightly Superior | 8 | 20 | 11
  Extremely Superior | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Vertical Lens Centration Grade After 4 Weeks of Comfilcon A Wear
Description: Number of Participants with Vertical lens centration after 4 weeks of comfilcon A wear graded on a scale of -2 to 2 ( -2= Extremely inferior, -1 slightly inferior, 0=optimum, 1=slightly superior, 2=extremely superior)
Time Frame: 4 weeks
Population: One subject discontinued after dispensing visit
Measure: Count of Participants; unit: Participants
Arm/Group | Comfilcon A Contact Lens
Number analyzed (Participants) | 54
Participants
  Extremely Inferior | 0
  Slightly Inferior | 9
  Optimum | 38
  Slightly Superior | 7
  Extremely Superior | 0

12. Secondary Outcome: Number of Participants With Vertical Lens Centration Grade
Description: as for outcome 10
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Contact Lens | Stenfilcon A Contact Lens
Number analyzed (Participants) | 51 | 52
Participants
  Extremely Inferior | 0 | 0
  Slightly Inferior | 10 | 4
  Optimum | 22 | 37
  Slightly Superior | 19 | 11
  Extremely Superior | 0 | 0

13. Secondary Outcome: Number of Participants With Lens Corneal Coverage Grade
Description: Number of Participants with Lens Corneal coverage graded on a scale -2 to 2 ( -2=extremely inadequate, -1=slightly inadequate, but acceptable, 0=optimum, 1=slightly excessive, but acceptable, 2=extremely excessive)
Time Frame: Baseline (after 5 minutes of lens dispense)
Measure: Count of Participants; unit: Participants
Arm/Group | Comfilcon A Contact Lens | Somofilcon A Contact Lens | Stenfilcon A Contact Lens
Number analyzed (Participants) | 55 | 51 | 53
Participants
  Extremely Inadequate | 0 | 0 | 0
  Slightly inadequate | 3 | 23 | 1
  Optimum | 48 | 26 | 46
  Slightly excessive | 4 | 2 | 6
  Extremely excessive | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Lens Corneal Coverage Grade After 4 Weeks of Comfilcon A Wear
Description: Number of Participants with Lens Corneal coverage after 4 weeks of comfilcon A wear graded on a scale -2 to 2 ( -2=extremely inadequate, -1=slightly inadequate, but acceptable, 0=optimum, 1=slightly excessive, but acceptable, 2=extremely excessive)
Time Frame: 4 weeks
Population: One subject discontinued after dispensing Visit
Measure: Count of Participants; unit: Participants
Arm/Group | Comfilcon A Contact Lens
Number analyzed (Participants) | 54
Participants
  Extremely Inadequate | 0
  Slightly inadequate | 4
  Optimum | 43
  Slightly excessive | 6
  Extremely excessive | 1

15. Secondary Outcome: Number of Participants With Lens Corneal Coverage Grade
Description: as for outcome 13
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Contact Lens | Stenfilcon A Contact Lens
Number analyzed (Participants) | 51 | 52
Participants
  Extremely Inadequate | 0 | 0
  Slightly inadequate | 20 | 3
  Optimum | 30 | 43
  Slightly excessive | 1 | 6
  Extremely excessive | 0 | 0

16. Secondary Outcome: Number of Participants With Post-Blink Movement Grade
Description: Number of Participants with Post-blink movement graded on a scale of -2 to 2 ( -2=extremely inadequate, -1=slightly inadequate, but acceptable, 0=optimum, 1=slightly excessive, but acceptable, 2=extremely excessive)
Time Frame: Baseline (after 5 minutes of lens dispense)
Measure: Count of Participants; unit: Participants
Arm/Group | Comfilcon A Contact Lens | Somofilcon A Contact Lens | Stenfilcon A Contact Lens
Number analyzed (Participants) | 55 | 51 | 53
Participants
  Extremely inadequate | 0 | 0 | 0
  Slightly inadequate | 11 | 6 | 7
  Optimum | 35 | 33 | 31
  Slightly excessive | 9 | 12 | 15
  Extremely excessive | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Post-Blink Movement Grade After 4 Weeks of Comfilcon A Wear
Description: Number of Participants with Post-blink movement after 4 weeks of comfilcon A wear graded on a scale of -2 to 2 ( -2=extremely inadequate, -1=slightly inadequate, but acceptable, 0=optimum, 1=slightly excessive, but acceptable, 2=extremely excessive)
Time Frame: 4 weeks
Population: One subject discontinued after dispensing visit
Measure: Count of Participants; unit: Participants
Arm/Group | Comfilcon A Contact Lens
Number analyzed (Participants) | 54
Participants
  Extremely inadequate | 0
  Slightly inadequate | 6
  Optimum | 38
  Slightly excessive | 10
  Extremely excessive | 0

18. Secondary Outcome: Number of Participants With Post-Blink Movement Grade
Description: as for outcome 16
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Contact Lens | Stenfilcon A Contact Lens
Number analyzed (Participants) | 51 | 52
Participants
  Extremely inadequate | 0 | 0
  Slightly inadequate | 5 | 5
  Optimum | 34 | 28
  Slightly excessive | 12 | 19
  Extremely excessive | 0 | 0

19. Secondary Outcome: Investigator Lens Fit Acceptance
Description: Lens fit acceptance investigator rating for acceptable and optimum fits on 1-5 Likert Scale (1=strongly agree, 2- Agree. 3- Neither agree not disagree, 4- Disagree, 5=strongly disagree)
Time Frame: Baseline (after 5 minutes of lens dispense)
Measure: Number; unit: percentage of lenses
Arm/Group | Comfilcon A Contact Lens | Somofilcon A Contact Lens | Stenfilcon A Contact Lens
Number analyzed (Participants) | 55 | 51 | 53
percentage of lenses
  Acceptable Fits | 100 | 100 | 100
  Optimum Fits | 27 | 16 | 28

20. Secondary Outcome: Investigator Lens Fit Acceptance for Comfilcon A After 4 Weeks of Use
Description: Lens fit acceptance investigator rating for comfilcon A after 4 weeks of use for acceptable and optimum fits on 1-5 Likert Scale (1=strongly agree, 2- Agree. 3- Neither agree not disagree, 4- Disagree, 5=strongly disagree)
Time Frame: 4 weeks
Population: One subject discontinued after dispensing visit
Measure: Number; unit: percentage of lenses
Arm/Group | Comfilcon A Contact Lens
Number analyzed (Participants) | 54
percentage of lenses
  Acceptable Fits | 98
  Optimum Fits | 33

21. Secondary Outcome: Investigator Lens Fit Acceptance
Description: as for outcome 19
Time Frame: 1 week
Measure: Number; unit: percentage of lenses
Arm/Group | Somofilcon A Contact Lens | Stenfilcon A Contact Lens
Number analyzed (Participants) | 51 | 52
percentage of lenses
  Acceptable Fits | 100 | 100
  Optimum Fits | 10 | 21

ADVERSE EVENTS:
Time Frame: From dispense up to 4 weeks for comfilcon A contact lens and from dispense up to one week for somofilcon A and stenfilcon A contact lens, up to 6 weeks total.
Description: Two subjects discontinued from somofilcon A intervention after dispensing. 53 subjects were considered at risk for adverse events for Somofilcon A Contact Lens Arm/Group..
Groups:
- Comfilcon A Contact Lens: All participants were fitted to wear comfilcon A lens on a daily wear, reusable basis for 1 month.
  comfilcon A: Contact Lens
Arm/Group | Comfilcon A Contact Lens | Somofilcon A Contact Lens | Stenfilcon A Contact Lens
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/53 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/53 | 0/53
Other Adverse Events (participants affected / at risk) | 0/55 | 0/53 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT04005885/Prot_SAP_000.pdf